CLINICAL TRIAL: NCT02618525
Title: Comparison of the Supraorbital Pressure and Jaw Thrust as Indicators for Depth of Anesthesia for Laryngeal Mask Airway Insertion in Children
Brief Title: Supraorbital Pressure Versus Jaw Thrust for Assessing the Adequate Depth of Anesthesia for LMA Insertion in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Asish Subedi, Principal Investigator, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Acd/10/071/072
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supraorbital pressure (Active Comparator): Supraorbital pressure is applied by applying pressure over the notch on the inner aspect of eyebrow.
  Interventions: Other: Jaw thrust maneuver
- Jaw thrust maneuver (Active Comparator): Jaw thrust maneuver is performed by placing the index and middle fingers to physically pull the posterior aspects of the mandible upwards while their thumbs push down on the chin to open the mouth.
  Interventions: Other: Supraorbital pressure

INTERVENTIONS:
Other: Supraorbital pressure — Supraorbital pressure is applied by applying pressure over the notch on the inner aspect of eyebrow.
  Arms: Jaw thrust maneuver
Other: Jaw thrust maneuver — Jaw thrust is performed by placing the index and middle fingers to physically pull the posterior aspects of the mandible upwards while their thumbs push down on the chin to open the mouth.
  Arms: Supraorbital pressure

SUMMARY:
BACKGROUND AND OBJECTIVES

The purpose of this study is to assess whether the loss of motor response to supraorbital pressure can be an alternative to that of jaw thrust to predict optimal condition for laryngeal mask airway (LMA) insertion in children.

METHODOLOGY

Fifty children (ASA I-II), aged 2 to 10 years, scheduled to receive general anesthesia that required LMA insertion were randomized to receive either supraorbital pressure (SOP) (n = 25) or jaw thrust (JT) (n = 25), after the loss of verbal response and body movements with a standard anesthetic. When motor response to the study intervention was absent, the LMA was inserted.

DETAILED DESCRIPTION:
The investigators enrolled fifty consecutive participants (aged one to ten years) with ASA physical status I or II scheduled to receive general anesthesia for various surgical procedures. Participants were allowed to have solid food, formula milk or cow's milk up to six hours, mother's milk up to four hours and clear fluid up to two hours before surgery.

On reaching the pre-operative room, when the participant was still on mothers lap or on the bed baseline measurements of non-invasive blood pressure (NIBP), pulse oximeter (SpO2) and electrocardiography (ECG) were taken. Fifteen minutes before induction of anesthesia, all participants were premedicated with ketamine, either 4mg/kg intramuscularly into the gluteal region with 26 G needle, or with 0.5mg/kg intravenously if intravenous (IV) cannula was in place.

Devices for ECG, SpO2 and NIBP monitoring were attached to the participant after arrival in the operating room. IV line was then inserted, if not already present. Pre-oxygenation was done with 100% oxygen using an appropriate size face mask. Anesthesia was induced with IV fentanyl (2mcg/kg), and propofol (2-4 mg/kg) until the loss of response to verbal contact or loss of eyelash reflex. Spontaneous ventilation was first assisted and then controlled manually to maintain an end-tidal carbon dioxide partial pressure of 33-40 mmHg. No neuromuscular blocking agent was administered.

Supraorbital pressure or jaw thrust was performed after loss of response to verbal contact, or absence of body movements. In group SOP, supraorbital pressure was applied over the supraorbital notch for five seconds. In group JT, the jaw thrust was applied gently by lifting the angles of the mandible vertically upward for five seconds. An IV bolus dose of propofol (1 mg/kg) was added if there was a motor response to the supraorbital pressure or the jaw thrust and the test was repeated after ten seconds. A second bolus dose of propofol was repeated if positive motor response was still present. A negative physical response to the test was considered as the end point of induction to perform LMA insertion. A classic LMA of appropriate size was inserted immediately. Ease of insertion and mouth opening, development of coughing, swallowing, movement, laryngospasm, or gross purposeful movements during or within one minute of LMA insertion and additional dosage of propofol if required were recorded. The LMA insertion was considered unsuccessful if LMA could not be inserted after administration of second bolus dose of propofol. The number of attempts and the insertion conditions were recorded using a six variable three points scoring system(31)

* Mouth opening: 1 - Full, 2 - Partial (not ideal but permits easy opening of mouth), 3 - Nil
* Ease of LMA insertion 1 - Easy, 2 - Difficult, 3 - Impossible.
* Swallowing: 1 - Nil, 2 - Mild, 3 - Severe
* Coughing: 1 - Nil, 2 - Mild, 3 - Severe
* Laryngospasm: 1 - Nil, 2 - Mild (relieved by positive pressure ventilation), 3 - Severe (desaturation<90%)
* Movement: 1 - Nil, 2 - Mild (Finger) (some movement but did not affect positioning of LMA), 3 - Severe (Arm/leg) (holding of LMA was required and additional dose of induction agent given).

The investigators summed all the five scores to give a LMA insertion condition summed score which ranged from 0 to 12, a lower summed score indicating more favourable LMA insertion conditions.

Table: Laryngeal mask airway insertion score.

Variables 0 1 2

Mouth opening Complete Partial Impossible Ease of insertion Easy Difficult Impossible Swallowing Nil Partial Complete Coughing Nil Partial Complete Laryngospasm Nil Partial Complete Movement Nil Partial Gross

LMA cuff was inflated with air and was connected to Jackson-Rees modification of the Ayre's T-piece. Effective ventilation was determined by observing chest wall and bag movement, auscultation, and capnography.

Blood pressure, heart rate and percentage saturation of oxygen were recorded in the pre-operative room, immediately after LMA insertion, five, ten and fifteen minutes after LMA insertion.

Anesthesia was maintained with isoflurane in oxygen. After the closure of skin incision, removal of LMA was done when the participant was still in deep plane of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 and 2

Exclusion Criteria:

* Congenital, acute or chronic heart and lung disease, Skull fracture or orbital fracture

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of successful LMA insertion at first attempt | Upto 1 minute after LMA insertion

SECONDARY OUTCOMES:
Ease of insertion of LMA | Upto 1 minute after LMA insertion
Adequacy of mouth opening | Upto 1 minute after LMA insertion
Incidence of swallowing | Upto 1 minute after LMA insertion
Incidence of coughing | Upto 1 minute after LMA insertion
Incidence of laryngospasm | Upto 1 minute after LMA insertion
Incidence of movement | Upto 1 minute after LMA insertion
Additional bolus dose of propofol if required | Upto 1 minute after LMA insertion
LMA insertion score | Upto 1 minute after LMA insertion
Heart rate | Upto 5 minute after LMA insertion
Non invasive blood pressure | Upto 5 minute after LMA insertion

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Pokharel, MD, Study Director — B.P. Koirala Institute of Health Sciences; Asish Subedi, MD, Study Director — B.P. Koirala Institute of Health Sciences
Locations (1):
- B. P. Koirala Institute Of Health Sciences, Dharān, Nepal